CLINICAL TRIAL: NCT00025350
Title: A Randomized Phase II Trial of Two Dose Levels of ZD1839 (Iressa) (NSC 715055, IND 61187) in Patients With Recurrent Colorectal Adenocarcinoma
Brief Title: Gefitinib in Treating Patients With Recurrent Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000068952; E-6200
Record Dates: First submitted 2001-10-11; First posted 2003-10-22 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2006-01

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of recurrent metastatic colorectal cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of two different doses of gefitinib in treating patients who have recurrent metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 4-month progression-free survival rate in patients with recurrent metastatic colorectal adenocarcinoma treated with gefitinib.
* Determine the objective tumor response rate, progression, and overall survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a randomized, double-blind study. Patients are stratified according to ECOG performance status (0-1 vs 2), baseline serum CEA (less than 5 mg/L vs at least 5 mg/L), and number of metastatic sites (1 vs 2 or more). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral gefitinib once daily (twice daily on day 1 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive a higher dose of oral gefitinib as in arm I. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven adenocarcinoma of the colon or rectum
* Measurable disease
* Evidence of new or progressive metastatic disease within 6 months of last treatment
* Must have received prior systemic treatment with fluorouracil (and/or its analogs, with or without leucovorin calcium or levamisole) and irinotecan in the adjuvant or metastatic setting
* Metastatic tumor site accessible for biopsy
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN (5 times ULN if tumor involvement of the liver)

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing active or uncontrolled infections
* Other prior malignancies allowed provided prior therapy is discontinued and no evidence of disease
* No other uncontrolled illness or psychiatric illness/social situations that would preclude study
* Must be able to take and retain oral medications

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior signal transduction inhibitors (e.g., vascular endothelial growth factor-, vascular endothelial growth factor receptor-, and epidermal growth factor receptor-targeted agents) for colorectal cancer

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* No other prior cytotoxic chemotherapy (e.g., oxaliplatin) for colorectal cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No other prior systemic therapy for colorectal cancer
* No other prior investigational or approved agents for colorectal cancer
* No other concurrent investigational agents
* No concurrent antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mace L. Rothenberg, MD, FACP, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (16):
- United States (16):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Rothenberg ML, LaFleur B, Levy DE, Washington MK, Morgan-Meadows SL, Ramanathan RK, Berlin JD, Benson AB 3rd, Coffey RJ. Randomized phase II trial of the clinical and biological effects of two dose levels of gefitinib in patients with recurrent colorectal adenocarcinoma. J Clin Oncol. 2005 Dec 20;23(36):9265-74. doi: 10.1200/JCO.2005.03.0536. PMID 16361624
- [Result] Rothenberg ML, Lafleur B, Washington MK, et al.: Changes in epidermal growth factor receptor signaling in serum and tumor biopsies obtained from patients with progressive metastatic colorectal cancer (MCRC) treated with gefitinib (ZD1839): an Eastern Cooperative Oncology Group study. [Abstract] J Clin Oncol 22 (Suppl 14): A-3000, 195s, 2004.